CLINICAL TRIAL: NCT06589349
Title: Effects of Kangaroo Care on Circadian Rhythm, Growth and Physiological Effects of Newborns Effect of Parameters on Breast Milk Cortisol Levels: Randomized Controlled Study
Brief Title: Effects of Kangaroo Care on Circadian Rhythm, Growth and Physiological Effects
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sibel Küçükoğlu (Other)
Collaborators: Health Institutes of Turkey (Other Government)
Responsible Party: Sponsor-Investigator, Sibel Küçükoğlu, Responsible researcher (Prof), Selcuk University
Organization: Selcuk University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SelcukUni2535
Record Dates: First submitted 2024-04-19; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Newborn; Vitality; Sleep; Preterm Labor; Care Pattern, Maternal
MeSH Terms: conditions — Obstetric Labor, Premature | interventions — Kangaroo-Mother Care Method

STUDY DESIGN:
Intervention Model Description: In the study, randomization will be done by stratifying according to type of nutrition (breast milk-formula milk) and week of gestation (28-31+6 32-37), as it may affect sleep. After the blocks are created, the groups included in the study will be randomly assigned to the layers with the letters A and B, using the random numbers table obtained in the computer environment (www.random.org). Which group the children included in the study will be included in will be determined by an independent statistician and will be given to the researcher in a sealed envelope
Who Masked: Investigator
Masking Description: The sample size of the study was calculated using the G power program. In the power analysis performed with the t test, one-way hypothesis, 0.80 effect size, 90% power, 0.05 significance level, assignment rate: 1, it was determined that a total of 56 preterm babies (Experiment: 28, Control: 28) would provide sufficient sample size.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- kangaroo care group (Experimental): Kangaroo care will be performed twice a day, in the morning and evening, for three days, between 10:00 in the morning and 22:00 in the evening, 1 hour after the treatment and care practices applied to the baby. To measure breast milk cortisol levels, breast milk samples will be collected by the researcher by expressing breast milk at 12.00 on the 1st, 2nd and 3rd days of the experimental and control groups.
  Interventions: Behavioral: Kangaroo Care
- Control Group (No Intervention): Babies in the control group will be followed routinely in an incubator/cotton. It will be monitored for 70 minutes without any procedure or application, and as in the experimental group, stimuli that will disturb the baby during this period will be tried to be controlled. If mothers in this group want to do kangaroo care, they will be encouraged, not prevented. However, mothers in this group who start giving kangaroo care at least twice a day for three days will be excluded from the study. To measure breast milk cortisol levels, samples of mothers in the control group will be collected by expressing breast milk at 12:00

INTERVENTIONS:
Behavioral: Kangaroo Care — Physiological parameters will be measured in the Day (10:00) - Night (22:00) cycle for 3 days, just before being taken into kangaroo care in the experimental group, and when the kangaroo care is terminated, the baby will be measured in the mother's arms. Then, the mother and baby will be placed in kangaroo care for a minimum of 70 minutes
  Arms: kangaroo care group

SUMMARY:
This study was planned to investigate the effect of premature babies receiving regular kangaroo care in the NICU on circadian rhythm, growth and physiological parameters, and breast milk cortisol levels

DETAILED DESCRIPTION:
Kangaroo Care (KC) may have positive effects on biological phase markers of immature circadian rhythms in newborns. KC provides circadian rhythm development by reducing the stress of newborns. Skin-to- skin contact intervention, which is similar to kangaroo care, affects the ẞ-endorphin concentration, which reduces pain in premature babies, and is known to reduce cortisol levels. KC, which supports exclusive breastfeeding and breastfeeding, can affect the circadian rhythm in newborns by providing information about the time of day to newborns through the increase in breastfeeding rates and the hormones and immune elements contained in breast milk. Although there are a limited number of studies in the literature examining the circadian rhythm or sleep-wake cycle of babies in the neonatal intensive care unit, no study has been found examining the circadian rhythm of babies receiving regular kangaroo care using brain imaging methods. In this respect, the study has unique value. In addition, within the scope of the study, regular kangaroo care for three days had a positive effect on the growth and physiological parameters of babies any studies examining the effect of breast milk on cortisol levels No study was found.

ELIGIBILITY:
Inclusion Criteria:

* Being between 28+0-37 weeks of pregnancy,
* Birth weight >1000 g,
* APGAR score >7 at the 5th minute after birth,
* Ability to feed every 2-3 hours

Exclusion Criteria:

* Getting mechanical ventilation support
* Undergoing surgery
* Having diseases and disorders such as congenital brain malformations, meningitis, seizures, encephalopathy, congenital abnormalities, history of intraventricular bleeding, herpes, sepsis and heart or metabolic diseases.
* Taking medication that affects sleep patterns, such as theophylline, phenobarbital, midazolam, caffeine, fentalnil
* Having developed intraventricular hemorrhage

Ages: 28 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 56 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Newborn Circadian Rhythm Tracking Chart | First Day, (10:00-12:00 AM) - First Night (22:00- 24:00 PM)
  To measure circadian rhythms, BIS spectrometry will be attached to the baby's forehead area, as specified in the user manual, after the babies in the experimental and control groups are given group care in the morning and evening
  The device provides a different application to babies as it records the duration of being in "awake, REM, N-REM/ STAGE I, N-REM/ STAGE II, N-REM/ STAGE III, N-REM/ STAGE IV" measured in 5-minute periods. It will not be done. The sensor will be removed from the baby's forehead at the next care hour. At the end of 3 days, records will be taken from the BIS monitor and recorded in the "Newborn Circadian Rhythm Tracking Chart
Breast milk cortisol levels Tracking Chart | First Day (12:00AM) - first Night (24:00 PM)
  To measure breast milk cortisol levels, breast milk samples will be collected by the researcher by expressing breast milk at 12.00 on the 1st, 2nd and 3rd days of the experimental and control groups. This period was determined by considering the possibility of terminating kangaroo care in the experimental group as it coincided with the babies' care and feeding hours at 12:00, and the times when the mother would want to receive kangaroo care for more than 70 minutes, and the maximum kangaroo care would last 120 minutes
Growth Tracking Chart | First Day (10:00 AM)
  The chart was created by the researcher in such a way that body weight (g) from growth parameters would be recorded daily for 3 days.
Physiological Parameter Follow-up Form- body temperature (°C) | First Day (10:00 AM) and First Night (22:00 PM)
  Body temperature (°C) found in the Physiological Parameter Follow-up Form will be measured at 10:00 and 22:00 on the first day.
Physiological Parameter Follow-up Form-oxygen saturation (mmHg) | First Day (10:00 AM) and First Night (22:00 PM)
  Oxygen saturation found in the Physiological Parameter Follow-up Form will be measured at 10:00 and 22:00 on the first day.
Physiological Parameter Follow-up Form-heart rate (min) | First Day (10:00AM) and First Night (22:00 PM)
  Heart rate found in the Physiological Parameter Follow-up Form will be measured at 10:00 and 22:00 on the first day.
Physiological Parameter Follow-up Form-respiratory rate (min) | First Day (10:00 AM) and First Night (22:00 PM)
  Respiratory rate found in the Physiological Parameter Follow-up Form will be measured at 10:00 and 22:00 on the first day.

SECONDARY OUTCOMES:
Newborn Circadian Rhythm Tracking Chart | Second Day (10:00-12:00 AM) - Second Night (22:00-24:00 PM)
  To measure circadian rhythms, BIS spectrometry will be attached to the baby's forehead area, as specified in the user manual, after the babies in the experimental and control groups are given group care in the morning and evening
  The device provides a different application to babies as it records the duration of being in "awake, REM, N-REM/ STAGE I, N-REM/ STAGE II, N-REM/ STAGE III, N-REM/ STAGE IV" measured in 5-minute periods. It will not be done. The sensor will be removed from the baby's forehead at the next care hour. At the end of 3 days, records will be taken from the BIS monitor and recorded in the "Newborn Circadian Rhythm Tracking Chart
Newborn Circadian Rhythm Tracking Chart | Third Day (10:00-12:00 AM) - Third Night (22:00-24:00 PM)
  To measure circadian rhythms, BIS spectrometry will be attached to the baby's forehead area, as specified in the user manual, after the babies in the experimental and control groups are given group care in the morning and evening
  The device provides a different application to babies as it records the duration of being in "awake, REM, N-REM/ STAGE I, N-REM/ STAGE II, N-REM/ STAGE III, N-REM/ STAGE IV" measured in 5-minute periods. It will not be done. The sensor will be removed from the baby's forehead at the next care hour. At the end of 3 days, records will be taken from the BIS monitor and recorded in the "Newborn Circadian Rhythm Tracking Chart
Breast milk cortisol levels Tracking Chart | Second Day (12:00 AM) - Second Night (24:00 PM)
  To measure breast milk cortisol levels, breast milk samples will be collected by the researcher by expressing breast milk at 12.00 on the 1st, 2nd and 3rd days of the experimental and control groups. This period was determined by considering the possibility of terminating kangaroo care in the experimental group as it coincided with the babies' care and feeding hours at 12:00, and the times when the mother would want to receive kangaroo care for more than 70 minutes, and the maximum kangaroo care would last 120 minutes
Breast milk cortisol levels Tracking Chart | Third Day (12:00 AM) - Third Night (24:00 PM)
  To measure breast milk cortisol levels, breast milk samples will be collected by the researcher by expressing breast milk at 12.00 on the 1st, 2nd and 3rd days of the experimental and control groups. This period was determined by considering the possibility of terminating kangaroo care in the experimental group as it coincided with the babies' care and feeding hours at 12:00, and the times when the mother would want to receive kangaroo care for more than 70 minutes, and the maximum kangaroo care would last 120 minutes
Growth Tracking Chart | Second Day (10:00)
  The chart was created by the researcher in such a way that body weight (g) from growth parameters would be recorded daily for 3 days.
Growth Tracking Chart | Third Day (10:00 AM)
  The chart was created by the researcher in such a way that body weight (g) from growth parameters would be recorded daily for 3 days.
Physiological Parameter Follow-up Form- body temperature (°C) | Second Day (10:00 AM) - Second Night (22:00 PM)
  Body temperature (°C) found in the Physiological Parameter Follow-up Form will be measured at 10:00 and 22:00 on the second day.
Physiological Parameter Follow-up Form-oxygen saturation (mmHg) | Second Day (10:00 AM) - Second Night (22:00 PM)
  Oxygen saturation found in the Physiological Parameter Follow-up Form will be measured at 10:00 and 22:00 on the second day.
Physiological Parameter Follow-up Form-heart rate (min) | Second Day (10:00 AM) - Second Night (22:00 PM)
  Heart rate found in the Physiological Parameter Follow-up Form will be measured at 10:00 and 22:00 on the second day.
Physiological Parameter Follow-up Form-respiratory rate (min) | Second Day (10:00 AM) - Second Night (22:00 PM)
  Respiratory rate found in the Physiological Parameter Follow-up Form will be measured at 10:00 and 22:00 on the second day.
Physiological Parameter Follow-up Form- body temperature (°C) | Third Day (10:00 AM) - Third Night (22:00 PM)
  Body temperature (°C) found in the Physiological Parameter Follow-up Form will be measured at 10:00 and 22:00 on the third day.
Physiological Parameter Follow-up Form-oxygen saturation (mmHg) | Third Day (10:00 AM) - Third Night (22:00 PM)
  Oxygen saturation found in the Physiological Parameter Follow-up Form will be measured at 10:00 and 22:00 on the third day.
Physiological Parameter Follow-up Form-heart rate (min) | Third Day (10:00 AM) - Third Night (22:00 PM)
  Heart rate found in the Physiological Parameter Follow-up Form will be measured at 10:00 and 22:00 on the third day.
Physiological Parameter Follow-up Form-respiratory rate (min) | Third Day (10:00 AM) - Third Night (22:00 PM)
  Respiratory rate found in the Physiological Parameter Follow-up Form will be measured at 10:00 and 22:00 on the third day.

CONTACTS AND LOCATIONS:
Overall Officials: Sibel Kucukoglu, Prof, Study Director — Selcuk University
Locations (1):
- Selcuk University, Konya, Selcuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It will be shared after the article is published

REFERENCES:
- [Background] Kucukoglu S, Yilmaz Kurt F, Aytekin Ozdemir A, Ozcan Z. The Effect of Kangaroo Care on Breastfeeding and Development in Preterm Neonates. J Pediatr Nurs. 2021 Sep-Oct;60:e31-e38. doi: 10.1016/j.pedn.2021.02.019. Epub 2021 Mar 6. PMID 33750645
- [Background] Lan HY, Yin T, Chen JL, Chang YC, Liaw JJ. Factors Associated With Preterm Infants' Circadian Sleep/Wake Patterns at the Hospital. Clin Nurs Res. 2019 May;28(4):456-472. doi: 10.1177/1054773817724960. Epub 2017 Aug 9. PMID 28793784
- [Background] Martin-Montero A, Gutierrez-Tobal GC, Gozal D, Barroso-Garcia V, Alvarez D, Del Campo F, Kheirandish-Gozal L, Hornero R. Bispectral Analysis of Heart Rate Variability to Characterize and Help Diagnose Pediatric Sleep Apnea. Entropy (Basel). 2021 Aug 6;23(8):1016. doi: 10.3390/e23081016. PMID 34441156
- [Result] Gebuza G, Kazmierczak M, Lenska K. The effects of kangaroo mother care and music listening on physiological parameters, oxygen saturation, crying, awake state and sleep in infants in NICU. J Matern Fetal Neonatal Med. 2022 Oct;35(19):3659-3669. doi: 10.1080/14767058.2020.1836619. Epub 2020 Oct 20. PMID 33081550